CLINICAL TRIAL: NCT00110227
Title: Tai Chi Mind-Body Therapy for Chronic Heart Failure
Acronym: NEXT-Heart
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004P000390; R01AT002454 (NIH)
Record Dates: First submitted 2005-05-04; First posted 2005-05-05 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure
Keywords: Complementary Therapies; Tai Chi
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi (Experimental): 12-week tai chi program
  Interventions: Behavioral: 12-week Tai Chi Program
- Heart Health Education (Active Comparator): 12-week attention control
  Interventions: Behavioral: 12-week Education Program

INTERVENTIONS:
Behavioral: 12-week Tai Chi Program — 24 tai chi sessions. 2 sessions/week for 12 weeks.
  Arms: Tai Chi
Behavioral: 12-week Education Program — 24 Educational sessions. 2 sessions/week for 12 weeks.
  Arms: Heart Health Education

SUMMARY:
The purpose of this study is to determine the effects of a tai chi exercise program on functional capacity and health-related quality of life in patients with chronic heart failure (HF). This study will also examine the way tai chi influences mental, physical, and social functioning.

DETAILED DESCRIPTION:
HF is a major public health problem in the United States, affecting approximately 5 million adults. Despite recent advances in pharmacologic therapy and technologic devices, HF is the most common reason for hospitalization among Medicare patients and is reaching epidemic proportions as the population ages. New and inexpensive interventions that can improve functional capacity and quality of life and can delay disease progression are needed. Tai chi is a popular mind-body exercise that is a potential treatment for heart disease. This exercise incorporates both gentle physical activity and meditation, and it may be particularly suited to frail patients with HF. This study will examine the effects of a tailored tai chi program on functional capacity and quality of life in patients with HF.

Participants will be randomly assigned to either a tai chi program or heart health education for 12 weeks. Participants in both groups will undergo a bicycle stress test at study entry and will receive weekly training sessions of their assigned intervention. Self-report scales and questionnaires will be used to assess participants at study start and at the end of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic HF
* Percentage of blood pumped from the left ventricle (ventricular ejection fraction) less than 40% for at least 1 year prior to study entry
* Stable medical regimen, defined as no major changes in medication, in the 3 months prior to study entry
* New York Heart Association Classification of Class I (no activity limitations), Class II (slight activity limitations), or Class III (marked activity limitations)
* English-speaking

Exclusion Criteria:

* Unstable angina, myocardial infarction, cardiac resynchronization, or major cardiac surgery within 3 months prior to study entry
* History of cardiac arrest or diagnosis of peripartum cardiomyopathy within 6 months prior to study entry
* Unstable ventricular arrhythmias or structural valvular disease
* Current participation in a conventional cardiac rehabilitation program
* Inability to perform a bicycle stress test at study entry
* Lower extremity amputation or other inability to walk due to conditions other than HF
* Severe cognitive dysfunction preventing informed consent and understanding of tai chi concept
* Current regular practice of tai chi
* Current participation in a tai chi pilot study or other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-09; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
HF-specific quality of life | baseline, midpoint, endpoint, 6mo
functional capacity | baseline and endpoint
Walking Test | baseline, midpoint, endpoint

SECONDARY OUTCOMES:
General quality of life | baseline, midpoint, endpoint, 6mo
mood and emotional status | baseline, midpoint, endpoint, 6mo
exercise self-efficacy | baseline, midpoint, endpoint, 6mo
sense of coherence | baseline, midpoint, endpoint, 6mo
utility assessment | baseline, midpoint, endpoint, 6mo
beliefs, attitudes, and expectations | baseline, midpoint, endpoint
physical activity level | baseline, midpoint, endpoint
perceived social support | baseline, midpoint, endpoint
neurohormonal status | baseline, midpoint, endpoint
autonomic tone, heart rate variability | baseline and endpoint
echocardiography | baseline and endpoint
costs and use of HF services | baseline and endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Russell S. Phillips, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School; Ellen P. McCarthy, PhD, Study Director — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lown Cardiovascular Center, Brookline, Massachusetts

REFERENCES:
- [Background] Yeh GY, Wood MJ, Lorell BH, Stevenson LW, Eisenberg DM, Wayne PM, Goldberger AL, Davis RB, Phillips RS. Effects of tai chi mind-body movement therapy on functional status and exercise capacity in patients with chronic heart failure: a randomized controlled trial. Am J Med. 2004 Oct 15;117(8):541-8. doi: 10.1016/j.amjmed.2004.04.016. PMID 15465501
- [Result] Yeh GY, McCarthy EP, Wayne PM, Stevenson LW, Wood MJ, Forman D, Davis RB, Phillips RS. Tai chi exercise in patients with chronic heart failure: a randomized clinical trial. Arch Intern Med. 2011 Apr 25;171(8):750-7. doi: 10.1001/archinternmed.2011.150. PMID 21518942